CLINICAL TRIAL: NCT01449162
Title: A Prospective, Multicenter, Randomised, Double-blind, Placebo-controlled, 2-parallel Groups, Phase 3 Study to Compare the Efficacy and the Safety of Masitinib at 6 mg/kg/Day Versus Placebo in the Treatment of Patients With Severe Persistent Asthma Treated With Oral Corticosteroids
Brief Title: Masitinib in Treatment of Patients With Severe Persistent Asthma Treated With Oral Corticosteroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB07015
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Asthma
Keywords: severe persistent asthma; tyrosine kinase inhibitor
MeSH Terms: conditions — Asthma | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Masitinib as add-on to oral corticosteroids (Experimental): Participants receive masitinib (6 mg/kg/day), given orally twice daily, as add-on to oral corticosteroids
  Interventions: Drug: Masitinib
- Placebo as add-on to oral corticosteroids (Placebo Comparator): Participants receive placebo (6 mg/kg/day), given orally twice daily, as add-on to oral corticosteroids
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Masitinib — 6 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib as add-on to oral corticosteroids
Drug: Placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo as add-on to oral corticosteroids

SUMMARY:
The study objective is to compare the efficacy and the safety of masitinib at 6 mg/kg/day versus placebo in the treatment of patients with Severe Persistent Asthma treated with oral corticosteroids.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor. It is known that activation of inflammatory cells, such as mast cells, and fibrous tissue remodeling are associated with c-Kit, Lyn and PDGFR kinase signaling pathways; all key targets of masitinib. The objective of this study is to compare the efficacy and safety of masitinib at 6 mg/kg/day versus matched placebo in severe persistent asthma patients that is uncontrolled with oral corticosteroids. The primary outcome measure will be severe asthma exacerbation rate over duration of the treatment.

ELIGIBILITY:
Main inclusion criteria:

1. Patient with severe asthma and already treated with oral corticosteroids at a minimal daily dose of 7.5 mg prednisone or equivalent for at least 3 months prior to screening visit
2. Patient treated with oral corticosteroids during at least one period of 21 days, from 1 year prior to screening to 3 months before screening
3. Patient with no significant change in the regular asthma medication, no severe asthma exacerbation for at least 4 weeks prior to screening visit
4. Non-smoker patient for at least 1 year and with a prior tobacco consumption < 10 packs/year

Main exclusion criteria:

1. Patient with active lung disease other than asthma (e.g. chronic bronchitis)
2. Female patient who is pregnant or lactating
3. Asthmatic patient still exposed to allergens or to triggering factors influencing asthma control
4. Patient with history of acute infectious sinusitis or respiratory tract infection within 4 weeks prior to screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Severe asthma exacerbation rate | Duration of patient treatment exposure, assessed until withdrawal from study, study completion date, or for a maximum of 60 months
  The number of severe asthma exacerbations over time frame of outcome measure

SECONDARY OUTCOMES:
Asthma exacerbation rate | Duration of patient treatment exposure, assessed until withdrawal from study, study completion date, or for a maximum of 60 months
  The number of asthma exacerbations over time frame of outcome measure
ACQ Score | 36 weeks
  Asthma Control Questionnaire (ACQ) Score

CONTACTS AND LOCATIONS:
Overall Officials: Lavinia Davidescu, MD, PhD, Principal Investigator — University of Medicine and Pharmacy Oradea, Oradea, Romania
Locations (8):
- Dr. Georgi Stranski University Hospital, Pleven, Bulgaria
- Hospital Polyclinic Melnik, Mělník, Czechia
- France (3):
  - Hospital La Cavale Blanche, Brest
  - l'Hopital Albert Calmette, Lille
  - l'Hopital de la Croix Rousse, Lyon
- University of Debrecen Medical and Health Science Center, Debrecen, Hungary
- King George Hospital, Hyderabad, India
- Hospital Universitario Doctor Peset, Valencia, Spain